CLINICAL TRIAL: NCT00664508
Title: Mobility Assessment of Patients With Total Hip Arthroplasty: Joint Mechanics and Rehabilitation
Brief Title: Mobility Assessment of Patients With Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2007-390
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis; Arthroplasty; Hip Replacement
Keywords: Arthroplasty; Hip Replacement; motion analysis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Comparative study with a control group
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lateral approach (Active Comparator): Lateral approach Intervention: Motion Analysis. Standard AP/Lateral x-rays of the hips, functional assessment questionnaires and 3D joint mechanic assessment at the Biomechanics Laboratory
  Interventions: Procedure: Motion analysis
- Anterior approach (Active Comparator): Anterior approach Intervention: Motion Analysis. Standard AP/Lateral x-rays of the hips, functional assessment questionnaires and 3D joint mechanic assessment at the Biomechanics Laboratory
  Interventions: Procedure: Motion analysis
- Posterior approach (Active Comparator): Posterior approach Intervention: Motion Analysis. Standard AP/Lateral x-rays of the hips, functional assessment questionnaires and 3D joint mechanic assessment at the Biomechanics Laboratory
  Interventions: Procedure: Motion analysis

INTERVENTIONS:
Procedure: Motion analysis — Motion analysis will be administered to each of the three groups: Lateral approach, anterior approach and posterior approach

SUMMARY:
The purpose of this study is to describe the 3D joint biomechanics of the lower extremities of patients having had a total hip replacement or hip resurfacing surgery as compared to a healthy age and weight matched control group during level walking, stair ascent and descent, and entering and exiting the front seat of a car.

DETAILED DESCRIPTION:
Much research has shown that patients are generally satisfied with pain relief in the months and years following a total hip replacement (THR) or hip resurfacing procedure. However, many express dissatisfaction with their ability to perform daily activities, a reduced walking ability and long-term lower extremity muscle weakness. Given the general lack of knowledge surrounding joint motion of the lower extremities in the THR population, there is a need to characterize the joint mechanics of people having undergone THR, so that interventions and rehabilitation strategies can be designed to reduce post-operative complications and improve mobility.

ELIGIBILITY:
Inclusion Criteria:

* 15 patients between the ages of 50 and 75 yrs having undergone a primary total hip replacement or hip resurfacing within 6 to 18 months of the study will participate, as well as an equal number of age, sex, height and weight matched healthy control participants.

Exclusion Criteria:

* Potential participants for the control group will be asked if they have had previous lower limb ailments or surgery, and if they have they will be excluded. Moreover, the THR participants cannot have had secondary hip replacement due to infection, revision surgery, or a concomitant surgical procedure (i.e., graft). Participants from both groups cannot have had any medical conditions which could affect physical movement such as a stroke.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Joint mechanics of people having undergone total hip replacement | 6-18 months post surgery
  3D joint mechanics of the lower extremities during level walking, stair ascent and descent, and entering and exiting the front seat of the car

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Beaule, MD, FRCSC, Principal Investigator — University of Ottawa / The Ottawa Hospital
Locations (1):
- OHRI, Ottawa, Ontario, Canada